CLINICAL TRIAL: NCT03860103
Title: Placental Insufficiency Microcirculation Quantification by Ultrafast Doppler: an Observational Prospective Study
Brief Title: Placental Insufficiency Microcirculation Quantification by Ultrafast Doppler (MICRODOPPLER PLACENTA)
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0049
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Preeclampsia and Intrauterine Growth Restriction
Keywords: microDoppler; placenta; preeclampsia; intrauterine growth restriction
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify fetuses small for their gestational-age who have reached their appropriate growth potential from growth-restricted fetuses due to placental insufficiency is uneasy. Intra Uterine Growth Restriction (IUGR) increases the risk for indicated preterm delivery, neonatal mortality and morbidity. Therefore, improving the knowledge of the placental perfusion is essential to better identify and manage fetal chronic oxygen deprivation associated with placental insufficiency. Thus, the investigators propose to study placental microcirculation with a more efficient Doppler than conventional Doppler use in clinical practice. The Ultrafast Doppler is being able to map placental blood flow and could have potential impact in placental insufficiency diagnosis and prevention. Moreover, this Doppler could discriminate maternal and fetal vascularization.

The hypothesis is that Ultrafast Doppler could help clinician to diagnose and manage preeclampsia and IUGR during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Patient who accepted to participate in the study
* Woman over 18 years old
* Affiliated to a social security scheme
* Mono-fetal pregnancy
* Patients with normal pregnancy between 11 and 42 weeks of amenorrhea
* Patients hospitalized for preeclampsia and / or intrauterine growth retardation, beyond 20 weeks of amenorrhea

Exclusion Criteria:

* Minors, adults under guardianship, protected persons
* Not affiliated to a social security scheme
* Multiple pregnancy

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Qualitative analysis (velocities) of intraplacental blood flow after acquisition of sequences in Ultrafast Doppler imaging | from the 12 week of gestation
Quantitative analysis (flow rates) of intraplacental blood flow after acquisition of sequences in Ultrafast Doppler | from the 12 week of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided